CLINICAL TRIAL: NCT04295876
Title: The BRIDGES Project: Bridging Resources to Engage Women in Integrated HIV Care and Support Services
Acronym: BRIDGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Stanford University (Other); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Jamila K. Stockman, Associate Professor, Vice Chief of Global Public Health, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 191314; HD15-SD-059 (Other Grant/Funding Number: California HIV/AIDS Research Program)
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: HIV/AIDS
Keywords: HIV Care Continuum; Ancillary Support Services
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Women assigned to the control arm will receive self-directed (non-PN supported) treatment as usual at the HIV care service provider of choice following the Ryan White standard of care (i.e., referrals to physical, dental and mental health services; case management; and ancillary services. Annual assessments (e.g., updates on insurance, housing, referrals needed, behavioral assessment [e.g., depression, substance use]) are conducted by a case manager. For women who have fallen out of care and re-engage care, case management begins with an interview and assessment of current needs. Goals are set to create an individual care plan related to medical care, housing, and other resources, as needed. Referrals are made to appropriate services (e.g., primary care, housing, benefits counseling, food, support services) based on the intake assessment.
- BRIDGES Arm (Experimental): Women assigned to The BRIDGES Project intervention arm will be connected with and receive Ryan White HIV/AIDS Program services (see above as described under Control Arm), as well as receive Peer Navigation support via one-on-one sessions, phone/text-based check-ins, and 6 unique syndemic-responsive 120 -minute group sessions designed to build coping skills (3 sessions) and assertive communication and behavior (3 sessions).
  Interventions: Behavioral: The BRIDGES Project Intervention

INTERVENTIONS:
Behavioral: The BRIDGES Project Intervention — The BRIDGES Project will use Peer Navigators, who are other women living with HIV who have had similar experiences and have been successful in accessing care, to help other women living with HIV to access HIV care and stay in HIV care. The BRIDGES Project will also provide support to women through group sessions co-facilitated by a licensed clinical therapist and Peer Navigator. Through participation in BRIDGES, women will: (1) build skills to cope with HIV care and treatment barriers (e.g., violence, trauma, adverse mental health, substance use); (2) be connected to HIV treatment and other support services (e.g., domestic violence, mental health, substance use); and (3) learn interpersonal skills to connect with support (e.g., service providers, peers, friends, family) when faced with new or ongoing barriers.
  Arms: BRIDGES Arm

SUMMARY:
The BRIDGES Project seeks to test a program intended to help women living with HIV who face specific barriers due to culture, gender, violence, trauma, adverse mental health, and substance use to be able to better access HIV care. This program was created and tried with women living with HIV, as previously studies have indicated that women with these experiences are less likely to have stable HIV care. The BRIDGES Project will use Peer Navigators, who are other women living with HIV who have had similar experiences and have been successful in accessing care, to help other women living with HIV to access HIV care and stay in HIV care. The BRIDGES Project will also provide support to women through group sessions co-facilitated by a licensed clinical therapist and Peer Navigator. Through participation in BRIDGES, women will: (1) build skills to cope with HIV care and treatment barriers (e.g., violence, trauma, adverse mental health, substance use); (2) be connected to HIV treatment and other support services (e.g., domestic violence, mental health, substance use); and (3) learn interpersonal skills to connect with support (e.g., service providers, peers, friends, family) when faced with new or ongoing barriers.

DETAILED DESCRIPTION:
The BRIDGES Project intervention is culturally-tailored intervention for syndemic-affected cis- and transgender women living with HIV/AIDS (WLHA) that aims to: 1) build skills to cope with syndemic-related affective distress, 2) facilitate linkages to both HIV treatment and relevant ancillary service providers (e.g., domestic violence, mental health, substance use), and 3) teach women interpersonal skills to activate social support networks (e.g., service providers, friends, family) when faced with new or ongoing barriers. Participants in the The BRIDGES Project are estimated to demonstrate improvements in HIV care outcomes (i.e., linkage to HIV care, self-efficacy in ART adherence, retention in HIV care) and syndemic-support outcomes (i.e., coping skills, activated social support networks, linkage to and receipt of ancillary support services) compared to HIV-infected women assigned to standard of care (self-guided access and use of Ryan White case management).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Identify as female, including cis-gender female or transgender female
* Living with HIV/AIDS
* Ability to speak and understand English
* Self-report one or more syndemic factor(s) [lifetime history of or current: trauma, physical violence and/or sexual violence, PTSD symptoms, substance use, adverse mental health]
* identification as one of the following: out-of-care or unstable in care, newly diagnosed, never in care, or linked to care but have fallen out of care]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender identifying
Enrollment: 24 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Linkage to Care | 3-months post-Baseline
  Documentation of a clinical visit date with an ART-prescribing provider (yes, no), assessed by medical record extraction; days to first clinical visit since baseline (continuous), assessed by medical record extraction
Linkage to Care | 6-months post-Baseline
  Documentation of a clinical visit date with an ART-prescribing provider (yes, no), assessed by medical record extraction; days to first clinical visit since baseline (continuous), assessed by medical record extraction
Self-Efficacy for ART Adherence | 3-months post-Baseline
  Validated self-report measures of ART regime adherence
Self-Efficacy for ART Adherence | 6-months post-Baseline
  Validated self-report measures of ART regime adherence
ART Initiation AND/OR Retention | 3-months post-Baseline
  Validated self-report measures of ART regime adherence
ART Initiation AND/OR Retention | 6-months post-Baseline
  Validated self-report measures of ART regime adherence
Retention in Care | 6-months post-Baseline
  2 clinic visits 90+days apart, or as directed by an ART prescribing provider, assessed by medical record extraction

SECONDARY OUTCOMES:
Coping Self-Efficacy | 6-months post-Baseline
  Validated Measure of Coping Self-Efficacy (Coping Self Efficacy, Chesney et al 2006; Scale of 1 to 10 where 10 is greater coping self-efficacy.)
Social Support Network Activation | 6-months post-Baseline
  Validated Measure of Social Support, (MMOS-SS; Moser et al. 2012; Scale of 1 to 5 where 5 is greater social support.)
Ancillary Support Service Linkage | 3-months post-Baseline
  Self-Reported Support Service Linkage
Ancillary Support Service Linkage | 6-months post-Baseline
  Self-Reported Support Service Linkage
Ancillary Support Service Access | 6-months post-Baseline
  Self-Reported Support Service Access

OTHER OUTCOMES:
ART Adherence | 6-months post-Baseline
  Validated self-report adherence measures, proportion of WLHA attaining HIV viral suppression (<200 copies/mL, assessed by medical record extraction).
ART Adherence | 12-months post-Baseline
  Validated self-report adherence measures, proportion of WLHA attaining HIV viral suppression (<200 copies/mL, assessed by medical record extraction).

CONTACTS AND LOCATIONS:
Overall Officials: Jamila K. Stockman, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Webster Building, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
No, sensitive research subject information with small population, could compromise anonymity of research subjects.